CLINICAL TRIAL: NCT01905982
Title: The Effect of Reflective Breathing Therapy Compared With Conventional Breathing Therapy on Dyspnoea, Activity and Parasympathetic Activities in Patients With COPD III-IV
Brief Title: The Effect of Reflective Breathing Therapy Compared With Conventional Breathing Therapy in Patients With Chronic Obstructive Pulmonary Disease (COPD) III-IV; part2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Head physician (department of pulmonology), Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RAT 2013; KBerchtesgadener
Record Dates: First submitted 2013-07-19; First posted 2013-07-23 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional breathing therapy (Experimental): first: conventional breathing therapy, second: reflectory breathing therapy
  Interventions: Procedure: conventional breathing therapy
- Reflectory breathing therapy (Experimental): first: Reflectory breathing therapy second:Conventional breathing therapy
  Interventions: Procedure: reflectory breathing therapy

INTERVENTIONS:
Procedure: reflectory breathing therapy — duration:2x60 minutes
  Arms: Reflectory breathing therapy
Procedure: conventional breathing therapy — duration:4x30 minutes
  Arms: Conventional breathing therapy

SUMMARY:
The purpose of this study is to determine whether different types of breathing therapies in patients with COPD III-IV decrease dyspnea, increase activity and have impact on parasympathetic activities.

ELIGIBILITY:
Inclusion Criteria:

* inpatient rehabilitation
* COPD (Gold stage III and IV)

Exclusion Criteria:

* severe exacerbation in the last four weeks
* acute infections
* fever
* neuritides
* severe osteoporosis
* skin disease
* manic depression

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change in BORG-Scale | Change from pre (minute 0) in Borg Scale and directly post intervention
  Instrument for self-reported dyspnea; modified BORG-scale ranges from 1 (no dyspnea) to 10 (maximum dyspnea)

SECONDARY OUTCOMES:
Change in lung volume | change from pre (minute0) in residual volume to post intervention
  measured by a bodyplethysmograph
physical activity | 48 h post intervention
  measured by Senswear
parasympathetic activities | baseline and post intervention
  measured via Biofeedback
Chronic Respiratory Questionnaire | baseline and post intervention
  health related quality of life
COPD Assessment Test | baseline and post intervention
  health related Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Prof. Dr., Study Chair — Schön Klinik Berchtesgadener Land; Tessa Schneeberger, Principal Investigator — Schön Klinik Berchtesgadener Land
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau, Bavaria, Germany